## Statistical analysis:

Statistical analysis is made by SPSS 18.0 software for Windows (IBM SPSS, NY). Continuous variables are compared by Student's t-test or the Mann-Whitney U test and SD (standard deviation) or the median and interquartile range. Categorical variables are compared using the chi-square test or Fisher's exact test. Logisrtic regression analysis is applied to assess the independent association between NAFLD and the prevalence of AF after adjustment for potential con-founders. A 2-tailed test and a P value less than 0.05 is considered statistically significant.